CLINICAL TRIAL: NCT03713437
Title: Measurement of Beta Cell Death in Individuals With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 0611-18-EP
Record Dates: First submitted 2018-10-15; First posted 2018-10-19 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Cystic Fibrosis-related Diabetes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Participants will provide serum sample to determine levels of fructosamine, interleukin 6, glutamic acid decarboxylase, insulin antibody, zinc transporter, IA-2 antibody, and differentially methylated insulin DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic Fibrosis: Serum sample will be drawn once
  Interventions: Diagnostic Test: Measurement of differentially methylated insulin DNA
- Healthy, age-matched controls: Serum sample will be drawn once
  Interventions: Diagnostic Test: Measurement of differentially methylated insulin DNA

INTERVENTIONS:
Diagnostic Test: Measurement of differentially methylated insulin DNA — A serum sample will be drawn to measure differentially methylated insulin DNA.

SUMMARY:
This study evaluates the feasibility of using differentially methylated insulin DNA, a biomarker of beta cell death, in determining the time course of beta cell death and development of diabetes in people with cystic fibrosis. Study participants with cystic fibrosis and healthy control participants will have a blood sample drawn in order to measure the levels of differentially methylated insulin DNA.

DETAILED DESCRIPTION:
Cystic fibrosis related diabetes (CFRD) causes increased morbidity and mortality in people with cystic fibrosis (CF). The prevalence of CFRD increases with age. While CFRD is diagnosed in only 2 percent of children under 10 year sof age, it is present in 19 percent of adolescents and up to 50 percent of adults with CF. Although CFRD is uncommon in children, recent animal and human studies have shown that milder glycemic abnormalities are common in infants and young children with CF. One of the proposed mechanisms for early glucose dysregulation in CF is related to ongoing beta cell death that may start at a very early age. The assay to be used in this study measures differentially methylated insulin DNA, released exclusively by beta cells, to determine levels of beta cell death. This assay has been shown to detect beta cell death in individuals at risk of developing type 1 diabetes. If this assay successfully detects beta cell death in individuals with CF, the investigators can identify critical time points of beta cell loss in people with CF. Understanding how and when glycemic dysregulation occurs in CF will lead to better treatment of CFRD in the future.

ELIGIBILITY:
Inclusion Criteria for Cystic Fibrosis Subjects:

* Age 0 - 21 years
* Diagnosis of CF by two CF-causing mutations or elevated sweat chloride test
* Normal glucose tolerance, impaired glucose tolerance, indeterminate glucose tolerance or CFRD
* Pancreatic insufficiency

Exclusion Criteria for Cystic Fibrosis Subjects:

* Age > 21 years
* Diagnosis of type 1 or type 2 diabetes
* Pregnancy
* Oral or IV steroid use in the past 2 weeks
* Pulmonary exacerbation requiring hospital admission in the past 2 weeks.
* Initiation of CFTR corrector or potentiator medication within 6 months

Inclusion Criteria for healthy, age-matched controls:

* Age 0 - 21 years

Exclusion Criteria for healthy, age-matched controls:

* Age > 21 years
* Diagnosis of type 1 or type 2 diabetes or pre-diabetes
* Disorders impacting pancreatic exocrine function
* Pregnancy
* Oral or IV steroid use in the past 2 weeks

Max Age: 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Subjects with CF between the age of 0 and 21 years who are at their baseline health and have not started CFTR modulator therapy within the past 6 months.
  Healthy, age-matched controls between 0 and 21 years of age who do not have pancreatic endocrine or exocrine dysfunction.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Levels of differentially methylated insulin DNA from infancy to early adulthood in people with cystic fibrosis | Level to be drawn once, usually within 3 months of recruitment into study.
  Levels of differentially methylated insulin DNA in people with CF from infancy to young adulthood will be measured and compared to levels in healthy, age-matched controls.

SECONDARY OUTCOMES:
Correlation between level of differentially methylated insulin DNA and oral glucose tolerance status in people with CF. | Level to be drawn once, usually within 3 months of recruitment into study.
  Levels of differentially methylated insulin DNA in adolescents and young adults with CF will be correlated with oral glucose tolerance status such as impaired glucose tolerance, indeterminate glucose tolerance and CFRD.
Correlation between level of differentially methylated insulin DNA and use of CFTR modulator therapy. | Level to be drawn once, usually within 3 months of recruitment into study.
  Measure differences in levels of differentially methylated insulin DNA in people with CF on CFTR modulator drugs and people with CF not on modulator therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley R Deschamp, MD, Principal Investigator — University of Nebraska
Locations (1):
- Children's Hospital and Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No